CLINICAL TRIAL: NCT02801734
Title: Pilot Trial of the Enhancing Quality of Life in Patients (EQUIP) Intervention for Patients With Advanced Lung Cancer
Brief Title: Enhancing Quality of Life in Patients (EQUIP) Intervention for Patients With Advanced Lung Cancer
Acronym: EQUIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCCSPG-YR2016-JAN-15
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Advanced Lung Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the EQUIP intervention group will individually receive four face-to-face sessions with a palliative care nurse.
  For all participants, whether in intervention or control, usual care is provided - the primary oncologist may make a referral for palliative care input if deemed appropriate.
  Interventions: Other: EQUIP
- Control (No Intervention): For all participants, whether in intervention or control, usual care is provided - the primary oncologist may make a referral for palliative care input if deemed appropriate.

INTERVENTIONS:
Other: EQUIP — Patients in the EQUIP intervention group will receive four face-to-face sessions. The focus of these sessions is to equip patients with the skills and strategies needed to cope with common symptoms experienced by lung cancer patients.
  Arms: Intervention

SUMMARY:
i. Project Background Patients with advanced lung cancer have a high symptom burden and low quality of life. Early palliative care improves patient outcomes in newly diagnosed advanced lung cancer patients, but previously tested models are not feasible for widespread adoption. Hence, the aim of this study is to pilot a more sustainable nurse-led intervention - Enhancing Quality of life in Patients (EQUIP).

ii. Hypothesis / Aim The aims of this study are three-fold. Firstly, the investigators aim to determine the feasibility and acceptability of the EQUIP intervention itself. Secondly, the investigators aim to obtain a tentative estimate of efficacy of the EQUIP intervention. Thirdly, the investigators aim to determine the data completion rate of patient reported outcome measures in the context of the EQUIP trial.

iii. Methods Patients with newly diagnosed stage 3 or stage 4 lung cancer will be recruited and randomized to the EQUIP intervention or usual care (control) group. Patients randomized to the EQUIP intervention group will receive four face-to-face sessions with a palliative care nurse. The content of these educational sessions will equip patients with the knowledge and skills to manage the three commonest symptoms of fatigue, breathlessness and anxiety.

All participants will complete the Functional Assessment of Cancer Therapy - Lung (FACT-L), the Hospital Anxiety and Depression Scale (HADS) and the stigma subscale at four time points: baseline, 4, 8 and 12 weeks after recruitment. Measures of healthcare use will also be recorded. Additionally, participants in the intervention group will complete a feedback survey after each intervention session.

A total sample of 60 patients (30 in each arm) will be recruited.

Clinical Significance

If successful, this study will lead to a larger scale phase III trial which tests various components of the EQUIP intervention, in order to develop a sustainable and effective model for the provision of palliative care to advanced lung cancer patients.

ELIGIBILITY:
Inclusion criteria

* Has stage 3 or 4 lung cancer
* ECOG 0,1 or 2
* Able and willing to participate in the EQUIP programme

Exclusion criteria

- Unable to communicate in English or Mandarin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks
  Patient quality of life will be measured by the Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire.
Quality of life | 8 weeks
  Patient quality of life will be measured by the Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire.
Quality of life | 12 weeks
  Patient quality of life will be measured by the Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire.
Psychological distress | 4 weeks
  Psychological distress will be measured by the Hospital Anxiety and Depression Scale (HADS).
Psychological distress | 8 weeks
  Psychological distress will be measured by the Hospital Anxiety and Depression Scale (HADS).
Psychological distress | 12 weeks
  Psychological distress will be measured by the Hospital Anxiety and Depression Scale (HADS).

SECONDARY OUTCOMES:
Number of participants with referral to palliative care services | 6 months
Number of hospital admissions | 6 months
Number of visits to the emergency department | 6 months

OTHER OUTCOMES:
Overall survival | 1 year
Number of participants who died at home | 1 year
Number of participants with anti-cancer therapy in the last 4 weeks of life | Last four weeks of life

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore